CLINICAL TRIAL: NCT01301768
Title: Nutritional Status of Iodine in the Pregnant Population of Catalonia: a Study of Dietary Habits and Urinary Iodine
Brief Title: Group Education to Improve the Iodine Nutrition in Pregnancy: Cluster Randomized Trial
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: the intervention could not be performed. All participants received Usual clinical practice
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Responsible Party: Principal Investigator, USR Metropolitana Nord, Tecnic de Recerca, Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PI071265
Record Dates: First submitted 2010-05-31; First posted 2011-02-23 (Estimated); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Dietary Intervention; Pregnancy Jail; Iodine Deficiency
Keywords: Dietary Intervention; Pregnancy Jail; Iodine Deficiency; Iodine Nutrition; Dietary Habits; Urinary Iodine; Pregnancy; Group Education; Cluster Randomized Trial; Primary Health Care
MeSH Terms: conditions — Feeding Behavior | interventions — Diet Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group Education (Experimental): Group educational workshops about dietary habits in the first trimester because it is when organogenesis occurs and therefore when the iodine deficiency in the mother is an important risk in the development of the fetal central nervous system.
  Interventions: Other: Group Education
- Usual care (No Intervention): Women in the control group receive the usual care during the pregnancy

INTERVENTIONS:
Other: Group Education — Group educational workshops about dietary habits in the first trimester because it is when organogenesis occurs and therefore when the iodine deficiency in the mother is an important risk in the development of the fetal central nervous system.
  Other Names: Dietary Intervention
  Arms: Group Education

SUMMARY:
The purpose of this study is to assess the effectiveness of individual education versus group education about dietary habits and iodine supplementation to decrease iodine deficiency in pregnant women

DETAILED DESCRIPTION:
BACKGROUND: It is a priority to achieve an adequate nutritional status of iodine during pregnancy since iodine deficiency in this population may have repercussions on the mother during both gestation and post partum as well as on the foetus, the neonate and the child at different ages. According to the WHO, iodine deficiency is the most frequent cause of mental retardation and irrreversible cerebral lesions around the world. However, few studies have been published on the nutritional status of iodine in the pregnant population within the Primary Care setting, a health care level which plays an essential role in the education and control of pregnant women.

AIMS: 1.- To know the hygiene-dietetic habits related to the intake of foods rich in iodine and smoking during pregnancy. 2.- To determine the prevalence of iodine deficiency and the factors associated with its appearance during pregnancy.

METHODS/DESIGN: We will perform a cluster randomised, controlled, multicentre trial. Randomisation unit: Primary Care Team. Study population: 898 pregnant women over the age of 17 years attending consultation to a midwife during the first trimester of pregnancy in the participating primary care centres. Outcome measures: consumption of iodine-rich foods and iodine deficiency. Points of assessment: each trimester of the gestation. Intervention: group education during the first trimester of gestation on healthy hygiene-dietetic habits and the importance of an adequate iodine nutritional status. Statistical analysis: descriptive analysis of all variables will be performed as well as multilevel logistic regression. All analyses will be done carried out on an intention to treat basis and will be fitted for potential confounding factors and variables of clinical importance.

DISCUSSION: Evidence of generalised iodine deficiency during pregnancy could lead to the promotion of interventions of prevention such as how to improve and intensify health care educational programmes for pregnant women.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant Women in the first trimester
* Over the age of 17
* Receive routine care in their respective health center

Exclusion Criteria:

* Pregnant women who are in the second or third trimester.
* Pregnant women with diagnostic of thyroid disease.
* Pregnant women who do not have a phone.
* Pregnant women with communication difficulties (cognitive or sensory deterioration, language barrier).
* Pregnant women who do not consent to participate in the study.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2008-11; Primary Completion 2011-06 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Iodine deficiency | 36 weeks of pregnancy
  Urinary iodine excretion below 150 µg/l
Iodine deficiency | 24 weeks of pregnancy
  Urinari iodine excretion below 150 µg/l

SECONDARY OUTCOMES:
Date of birth | At baseline
Smoking | First trimester of pregnancy (14 weeks)
  Categories: yes / no
Iodized salt consumption | First trimester of pregnancy (14 weeks)
  Categories: yes / no
Iodine supplementation consumption | First trimester of pregnancy
  Categories: yes / no
Education Level | At baseline
  Categories: can not read or write, incomplete primary, completed primary, completed secondary and university
Ethnicity | At baseline
Number of pregnancies finishes | At baseline
Number of premature births | At baseline
Number of abortions | At baseline
Number of live births | At baseline
Trimester of pregnancy | First trimester of pregnancy
  Categories: yes / no
Glasses of milk a day (number) | First trimester of pregnancy
Yogurt per week (number) | First trimester of pregnancy
Servings of cheese per week (number) | First trimester of pregnancy
Usual preparation of vegetables | First trimester of pregnancy
  Categories: raw, fried, grilled / baked, steamed and boiled
Use of water to boil vegetables | First trimester of pregnancy
  Categories: yes / no
Vegetable consumption per week (number) | First trimester of pregnancy
Fish consumption per week (number) | First trimester of pregnancy
Usual preparation of fish | First trimester of pregnancy
  Categories: raw, fried, grilled / baked, steamed and boiled
Canned tuna consumption per week (number) | First trimester of pregnancy
Canned sardines consumption per week (number) | First trimester of pregnancy
Meat consumption per week (number) | First trimester of pregnancy
Cold meat consumption per week (number) | First trimester of pregnancy
Eggs consumption per week (number) | First trimester or pregnancy
Fruit consumption per week (number) | First trimester of pregnancy
Nuts consumption per week (number) | First trimester of pregnancy
Potassium iodide consumption | First trimester of pregnancy
Smoking | Second trimester of pregnancy (wk 15-wk 27 )
  Categories: yes / no
Smoking | Third trimester of pregnancy (wk28-wk40)
  Categories: yes / no
Iodized salt consumption | Second trimester of pregnancy
  Categories: yes / no
Iodized salt consumption | Third trimester of pregnancy
  Categories: yes / no
Iodine supplementation consumption | Second trimester of pregnancy
  Categories: yes / no
Iodine supplementation consumption | Third trimester of pregnancy
  Categories: yes / no
Trimester of pregnancy | Second trimester of pregnancy
  Categories: yes / no
Trimester of pregnancy | Third trimester of pregnancy
  Categories: yes / no
Glasses of milk a day (number) | Second trimester of pregnancy
Glasses of milk a day (number) | Third trimester of pregnancy
Yogurt per week (number) | Second trimester of pregnancy
Yogurt per week (number) | Third trimester of pregnancy
Servings of cheese per week (number) | Second trimester of pregnancy
Servings of cheese per week (number) | Third trimester of pregnancy
Usual preparation of vegetables | Second trimester of pregnancy
  Categories: raw, fried, grilled / baked, steamed and boiled
Usual preparation of vegetables | Third trimester of pregnancy
  Categories: raw, fried, grilled / baked, steamed and boiled
Use of water to boil vegetables | Second trimester of pregnancy
  Categories: yes / no
Use of water to boil vegetables | Third trimester of pregnancy
  Categories: yes / no
Vegetable consumption per week (number) | Second trimester of pregnancy
Vegetable consumption per week (number) | Third trimester of pregnancy
Fish consumption per week (number) | Second trimester of pregnancy
Fish consumption per week (number) | Third trimester of pregnancy
Usual preparation of fish | Second trimester of pregnancy
  Categories: raw, fried, grilled / baked, steamed and boiled
Usual preparation of fish | Third trimester of pregnancy
  Categories: raw, fried, grilled / baked, steamed and boiled
Canned tuna consumption per week (number) | Second trimester of pregnancy
Canned tuna consumption per week (number) | Third trimester of pregnancy
Canned sardines consumption per week (number) | Second trimester of pregnancy
Canned sardines consumption per week (number) | Third trimester of pregnancy
Meat consumption per week (number) | Second trimester of pregnancy
Meat consumption per week (number) | Third trimester of pregnancy
Cold meat consumption per week (number) | Second trimester of pregnancy
Cold meat consumption per week (number) | Third trimester of pregnancy
Eggs consumption per week (number) | Second trimester or pregnancy
Eggs consumption per week (number) | Third trimester or pregnancy
Fruit consumption per week (number) | Second trimester of pregnancy
Fruit consumption per week (number) | Third trimester of pregnancy
Nuts consumption per week (number) | Second trimester of pregnancy
Nuts consumption per week (number) | Third trimester of pregnancy
Potassium iodide consumption | Second trimester of pregnancy
Potassium iodide consumption | Third trimester of pregnancy
Iodine deficiency | Baseline at first trimester of pregnancy
  Urinary iodine excretion below 150 µg/l

CONTACTS AND LOCATIONS:
Overall Officials: Maria Teresa Torres Costa, Midwife, Principal Investigator — Institut Català de la Salut (ICS)
Locations (1):
- IDIAP Jordi Gol, Barcelona, Spain

REFERENCES:
- [Derived] Prieto G, Torres MT, Frances L, Falguera G, Vila L, Manresa JM, Casamitjana R, Barrada JR, Acera A, Guix D, Torrent A, Grau J, Toran P; IODEGEST study group. Nutritional status of iodine in pregnant women in Catalonia (Spain): study on hygiene-dietetic habits and iodine in urine. BMC Pregnancy Childbirth. 2011 Mar 8;11:17. doi: 10.1186/1471-2393-11-17. PMID 21385426